CLINICAL TRIAL: NCT01872910
Title: Evaluation of the Acute Analgesic Efficacy of a Single Dose of LY3023703 in Patients With Postsurgical Dental Pain: A Parallel, Double-Blind, Randomized, Placebo and Positive Control Study
Brief Title: A Study of LY3023703 Testing Pain Relief After Wisdom Teeth Removal
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14852; I6H-MC-MCBC (Other: Eli Lilly and Company)
Record Dates: First submitted 2013-06-05; First posted 2013-06-07 (Estimated); Results first posted 2017-12-14 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Acute Pain
Keywords: Wisdom tooth extraction
MeSH Terms: conditions — Acute Pain | interventions — Celecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Part A: Single oral administration of placebo matching corresponding LY3023703 dose administered orally once as a capsule post dental surgery.
  Part B: Single oral administration of placebo matching corresponding LY3023703 administered orally once as a capsule, post dental surgery and post dialysate probe placement.
  Part B of this study assessed whether LY3023703 selectively inhibited the prostaglandin E(PGE) surge in the wound dialysate during the postoperative period.
  Interventions: Drug: Placebo
- 30 milligrams (mg) LY3023703 (Experimental): Part A: Single oral administration of 30 milligrams (mg) LY3023703 administered orally once as a 30-milligrams (mg) capsule post dental surgery.
  Part B: Single oral administration of 30 milligrams (mg) LY3023703 administered orally once as a 30-mg capsule, post dental surgery and post dialysate probe placement.
  Part B of this study assessed whether LY3023703 selectively inhibited the prostaglandin E(PGE) surge in the wound dialysate during the postoperative period.
  Interventions: Drug: LY3023703
- 400 mg Celecoxib (Active Comparator): Part A: Single oral administration of 400 mg celecoxib (Positive control) administered orally once as two 200-mg capsules post dental surgery (Positive control).
  Participants received two 200-mg celecoxib capsules during Pre-Part B.The purpose of Pre-Part B was to develop proficiency in the dialysate placement, collection, and maintenance techniques before moving to Part B.
  Celecoxib was not administered in Part B.
  Part B of this study assessed whether LY3023703 selectively inhibited the prostaglandin E(PGE) surge in the wound dialysate during the postoperative period.
  Interventions: Drug: Celecoxib

INTERVENTIONS:
Drug: Placebo — Administered orally
  Arms: Placebo
Drug: LY3023703 — Administered orally
  Other Names: LY3023703 phosphate
  Arms: 30 milligrams (mg) LY3023703
Drug: Celecoxib — Administered orally
  Arms: 400 mg Celecoxib

SUMMARY:
The main purpose of this study is to test if a single dose of LY3023703 relieves pain after wisdom teeth removal. The study will last about one week for each participant, not including screening.

ELIGIBILITY:
Inclusion Criteria:

* Have at least 2 third molars which are clinically indicated for extraction. At least 1 molar should be a mandibular third molar with partial or complete bony impaction
* Are overtly healthy as determined by medical history and limited physical examination

Exclusion Criteria:

* Have chronic pain [for example (e.g.), fibromyalgia] or are experiencing episodic pain not related to the wisdom teeth (e.g., migraine pain) that could affect pain measurements as judged by the investigator
* Have temporomandibular joint disease or other condition which could affect pain processing or sensation, affect recovery from dental surgery, or otherwise affect ability to assess pain signal, in the opinion of the investigator
* Have substantial anxiety regarding dental or medical procedures as measured by the Corah Dental Anxiety Scale
* Are currently using or have recently used drugs that may confound assessment of the inflammatory response or pain including, but not limited to, nonsteroidal anti-inflammatory drugs (NSAIDs), aspirin and other analgesics, antihistamines, steroids, antidepressants, attention-enhancing drugs, or herbal supplements

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 124 (Actual)
Dates: Start 2013-06; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized to treatment groups when their dental pain intensity post oral surgery was moderate (or severe) as reported on a categorical 4-point scale: 0 (absent) to 3 (severe) and were marked on a 100 millimeter (mm) straight line visual analog scale (VAS) with a pain score ≥40 mm: 0 mm (no pain) to 100 mm (worst pain imaginable).
Groups:
- Part A - LY3023703: LY3023703: Administered orally once as a 30-milligrams (mg) capsule post dental surgery.
- Part A - Celecoxib: Celecoxib: Administered orally once as two 200-mg capsules post dental surgery (Positive control).
- Part A - Placebo: Placebo: Administered orally once as a capsule post dental surgery.
- Part B - LY3023703: LY3023703: Administered orally once as a 30-mg capsule, post dental surgery and post dialysate probe placement.
- Part B - Placebo: Placebo: Administered orally once as a capsule, post dental surgery and post dialysate probe placement.
- Pre-Part B - Celecoxib: Celecoxib: Administered orally once as two 200-mg capsules, post dental surgery and post dialysate probe placement. Prior to Part B, there was a technique transfer and training conducted to allow the site to develop proficiency in dialysate placement, collection and maintenance techniques.
Period: Overall Study
Arm/Group | Part A - LY3023703 | Part A - Celecoxib | Part A - Placebo | Part B - LY3023703 | Part B - Placebo | Pre-Part B - Celecoxib
Started | 30 | 31 | 30 | 15 | 15 | 3
Received Any Study Drug | 30 | 31 | 30 | 15 | 15 | 3
Completed | 28 | 31 | 28 | 15 | 15 | 3
Not Completed | 2 | 0 | 2 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who received study drug.
Groups:
- Part A - LY3023703: LY3023703: Administered orally once as a 30-mg capsule post dental surgery.
- Pre-Part B - Celecoxib: Celecoxib: Administered orally once as two 200-mg capsules, post dental surgery and post dialysate probe placement.
- Total: Total of all reporting groups
Arm/Group | Part A - LY3023703 | Part A - Celecoxib | Part A - Placebo | Part B - LY3023703 | Part B - Placebo | Pre-Part B - Celecoxib | Total
Number analyzed (Participants) | 30 | 31 | 30 | 15 | 15 | 3 | 124
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.5 (3.4) | 22.9 (4.3) | 22.9 (3.5) | 22.3 (3.2) | 24.8 (2.6) | 24.3 (2.5) | 22.98 (3.593)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 19 | 16 | 10 | 11 | 2 | 75
  Male | 13 | 12 | 14 | 5 | 4 | 1 | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 10 | 11 | 10 | 6 | 1 | 47
  Not Hispanic or Latino | 21 | 21 | 19 | 5 | 9 | 2 | 77
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Asian | 2 | 3 | 0 | 0 | 1 | 0 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 1 | 0 | 0 | 0 | 3
  White | 24 | 24 | 23 | 14 | 13 | 3 | 101
  More than one race | 3 | 2 | 6 | 1 | 1 | 0 | 13
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 30 | 31 | 30 | 15 | 15 | 3 | 124
VAS Pain Score at Post-Surgery Pre-Randomization [Mean (Standard Deviation); unit: mm] — A100-mm straight line is presented to the participant, with anchors of 0 mm at one end (no pain) and 100 mm at the other end (worst pain imaginable). The participant marks the line at the point that corresponds with his or her perceived intensity of pain.
  mm | 69.7 (13.1) | 77.0 (13.7) | 70.5 (10.7) | 75.1 (13.0) | 67.0 (6.1) | 72.6 (12.9) | 72.7 (12.7)

OUTCOME MEASURES:

1. Primary Outcome: Part A: Weighted Mean Change From Baseline in Pain Intensity Over the First 8 Hours Post-Dose Using VAS
Description: Pain intensity was rated by the participant on a 100-mm VAS: 0 mm (no pain) and 100 mm (worst pain imaginable). The participant marked the line at the point that corresponded with his or her perception of pain. Weighted mean change from baseline was calculated as: [the area under the change in pain intensity versus time curve] / 8 hours (h). The baseline pain intensity was the pain assessment prior to dosing of study medication (0 h). Least Squares (LS) mean were calculated using a Bayesian analysis of covariance analysis (ANCOVA) adjusted for treatment as a fixed effect and baseline pain VAS as a continuous covariate. The measure of dispersion reported is 95% Credible Interval (CrI) not Confidence Interval (CI). A negative direction indicates a pain reduction from baseline.
Time Frame: 0 to 8 h post-dose
Population: Full Analysis Set (FAS): Part A participants who were randomly assigned to treatment who received at least 1 dose of study medication and who had at least 1 postdose efficacy assessment. Pain assessments after rescue medication were imputed using last observation carried forward (LOCF) from the pain assessment prior to rescue therapy.
Measure: Least Squares Mean (95% Confidence Interval); unit: mm
Arm/Group | Part A - LY3023703 | Part A - Celecoxib | Part A - Placebo
Number analyzed (Participants) | 30 | 31 | 30
mm | -3.8 [-11.4 to 4.0] | -47.4 [-55.2 to -39.4] | -12.7 [-20.6 to -4.8]
Statistical Analysis 1: Comparison: Part A - LY3023703 vs Part A - Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = 9.0, 95% CI 2-sided [-2.1 to 20.0] — 95% CrI is reported here, not the CI
Statistical Analysis 2: Comparison: Part A - Celecoxib vs Part A - Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = -34.6, 95% CI 2-sided [-45.7 to -23.2] — 95% CrI is reported here, not the CI
Statistical Analysis 3: Comparison: Part A - LY3023703 vs Part A - Celecoxib; Test type: Superiority or Other; Mean Difference (Final Values) = 43.6, 95% CI 2-sided [32.7 to 54.9] — 95% CrI is reported here, not the CI

2. Secondary Outcome: Total Pain Relief (TOPAR) Score at 4, 6, 8, 12 and 24 Hours Post-Dose
Description: TOPAR was calculated as the area under the pain relief versus time curve of the participant reported pain relief scores from the 5-point pain relief scale of 0 (no pain relief) to 4 (complete pain relief). LS mean were calculated using ANCOVA adjusted for treatment as a fixed effect. The measure of dispersion reported is CrI not CI. A negative direction indicated a pain relief from baseline.
  Pre-Part B used 3 participants in order for the study site to develop proficiency in the dialysate placement, collection, and maintenance techniques. There were no planned efficacy analysis for Pre-Part B per protocol.
Time Frame: 0 to 4, 0 to 6, 0 to 8, 0 to 12, and 0 to 24 h post-dose
Population: FAS: All data from all participants randomly assigned to treatment who received at least 1 dose of study medication and who had at least 1 post-dose efficacy assessment. Pain assessments after rescue medication were imputed using LOCF from the pain assessment prior to rescue therapy excluding Pre-Part B.
Measure: Least Squares Mean (95% Confidence Interval); unit: pain relief * h
Arm/Group | Part A - LY3023703 | Part A - Celecoxib | Part A - Placebo | Part B - LY3023703 | Part B - Placebo
Number analyzed (Participants) | 30 | 31 | 30 | 15 | 15
pain relief * h
  0 to 4 h | 2.2 [1.1 to 3.3] | 8.1 [7.0 to 9.2] | 3.6 [2.5 to 4.7] | 1.1 [-0.0 to 2.2] | 1.1 [-0.0 to 2.2]
  0 to 6 h | 3.8 [1.9 to 5.7] | 13.4 [11.5 to 15.2] | 6.3 [4.4 to 8.2] | 1.8 [-0.2 to 3.7] | 2.0 [0.1 to 3.9]
  0 to 8 h | 5.2 [2.5 to 8.0] | 18.4 [15.7 to 21.0] | 9.2 [6.5 to 12.0] | 2.3 [-0.5 to 5.1] | 3.1 [0.3 to 5.8]
  0 to 12 h | 8.3 [3.8 to 12.7] | 28.0 [23.6 to 32.3] | 15.1 [10.6 to 19.7] | 3.1 [-1.3 to 7.6] | 5.2 [0.7 to 9.6]
  0 to 24 h | 17.9 [7.8 to 27.9] | 57.3 [47.2 to 67.1] | 34.2 [24.2 to 44.2] | 5.4 [-4.8 to 15.8] | 12.4 [2.3 to 22.6]
Statistical Analysis 1: Comparison: Part A - LY3023703 vs Part A - Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = -1.3, 95% CI 2-sided [-2.9 to 0.2] — 95% CrI is reported here, not the CI. Estimation is for TOPAR 0 to 4 h
Statistical Analysis 2: Comparison: Part A - Celecoxib vs Part A - Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = 4.5, 95% CI 2-sided [2.9 to 6.0] — 95% CrI is reported here, not the CI. Estimation is for TOPAR 0 to 4 h
Statistical Analysis 3: Comparison: Part A - LY3023703 vs Part A - Celecoxib; Test type: Superiority or Other; Mean Difference (Final Values) = -5.9, 95% CI 2-sided [-7.4 to -4.3] — 95% CrI is reported here, not the CI. Estimation is for TOPAR 0 to 4 h
Statistical Analysis 4: Comparison: Part A - LY3023703 vs Part A - Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = -2.5, 95% CI 2-sided [-5.2 to 0.2] — 95% CrI is reported here, not the CI. Estimation is for TOPAR 0 to 6 h
Statistical Analysis 5: Comparison: Part A - Celecoxib vs Part A - Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = 7.1, 95% CI 2-sided [4.4 to 9.8] — 95% CrI is reported here, not the CI. Estimation is for TOPAR 0 to 6 h
Statistical Analysis 6: Comparison: Part A - LY3023703 vs Part A - Celecoxib; Test type: Superiority or Other; Mean Difference (Final Values) = -9.6, 95% CI 2-sided [-12.2 to -6.9] — 95% CrI is reported here, not the CI. Estimation is for TOPAR 0 to 6 h
Statistical Analysis 7: Comparison: Part A - LY3023703 vs Part A - Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = -4.0, 95% CI 2-sided [-7.9 to -0.1] — 95% CrI is reported here, not the CI. Estimation is for TOPAR 0 to 8 h
Statistical Analysis 8: Comparison: Part A - Celecoxib vs Part A - Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = 9.2, 95% CI 2-sided [5.3 to 13.0] — 95% CrI is reported here, not the CI. Estimation is for TOPAR 0 to 8 h
Statistical Analysis 9: Comparison: Part A - LY3023703 vs Part A - Celecoxib; Test type: Superiority or Other; Mean Difference (Final Values) = -13.1, 95% CI 2-sided [-16.9 to -9.3] — 95% CrI is reported here, not the CI. Estimation is for TOPAR 0 to 8 h
Statistical Analysis 10: Comparison: Part A - LY3023703 vs Part A - Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = -6.8, 95% CI 2-sided [-13.2 to 0.5] — 95% CrI is reported here, not the CI. Estimation is for TOPAR 0 to 12 h
Statistical Analysis 11: Comparison: Part A - Celecoxib vs Part A - Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = 12.9, 95% CI 2-sided [6.6 to 19.2] — 95% CrI is reported here, not the CI. Estimation is for TOPAR 0 to 12 h
Statistical Analysis 12: Comparison: Part A - LY3023703 vs Part A - Celecoxib; Test type: Superiority or Other; Mean Difference (Final Values) = -19.7, 95% CI 2-sided [-25.9 to -13.5] — 95% CrI is reported here, not the CI. Estimation is for TOPAR 0 to 12 h
Statistical Analysis 13: Comparison: Part A - LY3023703 vs Part A - Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = -16.3, 95% CI 2-sided [-30.8 to -2.0] — 95% CrI is reported here, not the CI. Estimation is for TOPAR 0 to 24 h
Statistical Analysis 14: Comparison: Part A - Celecoxib vs Part A - Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = 23.1, 95% CI 2-sided [9.0 to 37.2] — 95% CrI is reported here, not the CI. Estimation is for TOPAR 0 to 24 h
Statistical Analysis 15: Comparison: Part A - LY3023703 vs Part A - Celecoxib; Test type: Superiority or Other; Mean Difference (Final Values) = -39.4, 95% CI 2-sided [-53.2 to -25.3] — 95% CrI is reported here, not the CI. Estimation is for TOPAR 0 to 24 h
Statistical Analysis 16: Comparison: Part B - LY3023703 vs Part B - Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-1.5 to 1.6] — 95% CrI is reported here, not the CI. Estimation is for TOPAR 0 to 4 h
Statistical Analysis 17: Comparison: Part B - LY3023703 vs Part B - Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-2.9 to 2.4] — 95% CrI is reported here, not the CI. Estimation is for TOPAR 0 to 6 h
Statistical Analysis 18: Comparison: Part B - LY3023703 vs Part B - Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-4.7 to 3.1] — 95% CrI is reported here, not the CI. Estimation is for TOPAR 0 to 8 h
Statistical Analysis 19: Comparison: Part B - LY3023703 vs Part B - Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = -2.1, 95% CI 2-sided [-8.3 to 4.1] — 95% CrI is reported here, not the CI. Estimation is for TOPAR 0 to 12 h
Statistical Analysis 20: Comparison: Part B - LY3023703 vs Part B - Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = -7.0, 95% CI 2-sided [-21.4 to 7.6] — 95% CrI is reported here, not the CI. Estimation is for TOPAR 0 to 24 h

3. Secondary Outcome: Weighted Mean Change From Baseline in Pain Intensity Over the First 24 Hours Post-Dose as Measured by VAS
Description: Pain intensity was rated by the participant on a 100-mm VAS: 0 mm (no pain) and 100 mm (worst pain imaginable). The participant marked the line at the point that corresponded with his or her perception of post oral surgery pain. Weighted mean change from baseline was calculated as: [area under the change in pain intensity versus time curve] / [time period that is (i.e.) 24 h for 0 to 24 h endpoint]. The baseline pain intensity was the pain assessment prior to dosing of study medication. LS mean were calculated using ANCOVA adjusted for treatment, time and interaction of treatment as a fixed effect and baseline pain VAS as a continuous covariate. The measure of dispersion reported is the 95% CrI not CI. A negative direction indicated a pain reduction from baseline.
  Pre-Part B used 3 participants in order for the study site to develop proficiency in the dialysate placement, collection, and maintenance techniques. There were no planned efficacy analysis for Pre-Part B per protocol.
Time Frame: Part A and B: 0 to 4, 0 to 6, 0 to 12, and 0 to 24 h post-dose and Part B 0 to 8 h post-dose
Population: FAS: All data from all participants randomly assigned to treatment who received at least 1 dose of study medication and who had at least 1 post-dose efficacy assessment. Pain assessments after rescue medication were imputed using LOCF from the pain assessment prior to rescue therapy.
Measure: Least Squares Mean (95% Confidence Interval); unit: mm
Arm/Group | Part A - LY3023703 | Part A - Celecoxib | Part A - Placebo | Part B - LY3023703 | Part B - Placebo
Number analyzed (Participants) | 30 | 31 | 30 | 15 | 15
mm
  0 to 4 h | -3.2 [-9.7 to 3.2] | -40.5 [-47.0 to -33.8] | -8.5 [-15.1 to -1.6] | 1.0 [-6.9 to 9.1] | -0.6 [-8.5 to 7.5]
  0 to 6 h | -3.6 [-10.9 to 3.5] | -46.1 [-53.4 to -38.7] | -10.9 [-18.3 to -3.7] | 1.7 [-7.8 to 11.1] | -1.8 [-11.3 to 7.7]
  0 to 8 h | NA [NA to NA] — Part A results are contained in Outcome Measure 1. | NA [NA to NA] — Part A results are contained in Outcome Measure 1. | NA [NA to NA] — Part A results are contained in Outcome Measure 1. | 2.1 [-8.1 to 12.4] | -2.3 [-12.4 to 7.9]
  0 to 12 h | -4.0 [-12.4 to 4.7] | -47.5 [-56.1 to -38.8] | -14.7 [-23.2 to -6.1] | 1.0 [-6.9 to 9.1] | -0.6 [-8.5 to 7.5]
  0 to 24 h | -5.2 [-15.2 to 4.6] | -47.9 [-57.4 to -38.2] | -17.7 [-27.5 to -8.0] | 3.9 [-7.8 to 15.5] | -4.0 [-15.6 to 7.5]
Statistical Analysis 1: Comparison: Part A - LY3023703 vs Part A - Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = 5.3, 95% CI 2-sided [-4.2 to 14.5] — 95% CrI is reported here, not the CI. Estimation is for weighted mean change from baseline pain intensity for 0 to 4 h
Statistical Analysis 2: Comparison: Part A - Celecoxib vs Part A - Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = -32.0, 95% CI 2-sided [-41.5 to -22.4] — 95% CrI is reported here, not the CI. Estimation is for weighted mean change from baseline pain intensity for 0 to 4 h
Statistical Analysis 3: Comparison: Part A - LY3023703 vs Part A - Celecoxib; Test type: Superiority or Other; Mean Difference (Final Values) = 37.3, 95% CI 2-sided [27.8 to 46.5] — 95% CrI is reported here, not the CI. Estimation is for weighted mean change from baseline pain intensity for 0 to 4 h
Statistical Analysis 4: Comparison: Part A - LY3023703 vs Part A - Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = 7.3, 95% CI 2-sided [-2.9 to 17.6] — 95% CrI is reported here, not the CI. Estimation is for weighted mean change from baseline pain intensity for 0 to 6 h
Statistical Analysis 5: Comparison: Part A - Celecoxib vs Part A - Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = -35.1, 95% CI 2-sided [-45.6 to -24.6] — 95% CrI is reported here, not the CI. Estimation is for weighted mean change from baseline pain intensity for 0 to 6 h
Statistical Analysis 6: Comparison: Part A - LY3023703 vs Part A - Celecoxib; Test type: Superiority or Other; Mean Difference (Final Values) = 42.5, 95% CI 2-sided [32.1 to 52.7] — 95% CrI is reported here, not the CI. Estimation is for weighted mean change from baseline pain intensity for 0 to 6 h
Statistical Analysis 7: Comparison: Part A - LY3023703 vs Part A - Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = 10.7, 95% CI 2-sided [-1.0 to 23.0] — 95% CrI is reported here, not the CI. Estimation is for weighted mean change from baseline pain intensity for 0 to 12 h
Statistical Analysis 8: Comparison: Part A - Celecoxib vs Part A - Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = -32.7, 95% CI 2-sided [-45.1 to -20.3] — 95% CrI is reported here, not the CI. Estimation is for weighted mean change from baseline pain intensity for 0 to 12 h
Statistical Analysis 9: Comparison: Part A - LY3023703 vs Part A - Celecoxib; Test type: Superiority or Other; Mean Difference (Final Values) = 43.5, 95% CI 2-sided [31.3 to 55.5] — 95% CrI is reported here, not the CI. Estimation is for weighted mean change from baseline pain intensity for 0 to 12 h
Statistical Analysis 10: Comparison: Part A - LY3023703 vs Part A - Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = 12.4, 95% CI 2-sided [-1.6 to 26.2] — 95% CrI is reported here, not the CI. Estimation is for weighted mean change from baseline pain intensity for 0 to 24 h
Statistical Analysis 11: Comparison: Part A - Celecoxib vs Part A - Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = -30.2, 95% CI 2-sided [-44.0 to -16.0] — 95% CrI is reported here, not the CI. Estimation is for weighted mean change from baseline pain intensity for 0 to 24 h
Statistical Analysis 12: Comparison: Part A - LY3023703 vs Part A - Celecoxib; Test type: Superiority or Other; Mean Difference (Final Values) = 42.6, 95% CI 2-sided [28.6 to 56.5] — 95% CrI is reported here, not the CI. Estimation is for weighted mean change from baseline pain intensity for 0 to 24 h
Statistical Analysis 13: Comparison: Part B - LY3023703 vs Part B - Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = 1.6, 95% CI 2-sided [-9.7 to 12.9] — 95% CrI is reported here, not the CI. Estimation is for weighted mean change from baseline pain intensity for 0 to 4 h
Statistical Analysis 14: Comparison: Part B - LY3023703 vs Part B - Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = 3.5, 95% CI 2-sided [-9.8 to 16.8] — 95% CrI is reported here, not the CI. Estimation is for weighted mean change from baseline pain intensity for 0 to 6 h
Statistical Analysis 15: Comparison: Part B - LY3023703 vs Part B - Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = 4.5, 95% CI 2-sided [-9.9 to 19.0] — 95% CrI is reported here, not the CI. Estimation is for weighted mean change from baseline pain intensity for 0 to 8 h
Statistical Analysis 16: Comparison: Part B - LY3023703 vs Part B - Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = 5.9, 95% CI 2-sided [-9.2 to 21.1] — 95% CrI is reported here, not the CI. Estimation is for weighted mean change from baseline pain intensity for 0 to 12 h
Statistical Analysis 17: Comparison: Part B - LY3023703 vs Part B - Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = 7.8, 95% CI 2-sided [-8.4 to 24.2] — 95% CrI is reported here, not the CI. Estimation is for weighted mean change from baseline pain intensity for 0 to 24 h

4. Secondary Outcome: Summed Pain Intensity Difference (SPID) Over the First 24 Hours Post-Dose as Measured by a 4-point Categorical Scale
Description: The summed (time-weighted) pain intensity difference to baseline (SPID) at 4, 6, 8, 12, and 24 h post-dosing, as measured by a participant-rated 4-point categorical scale of 0 (no pain) to 3 (severe pain) and was calculated as: the area under the change in pain intensity versus time curve. Total scores range: -24 (best) to 8 (worst) for SPID 0 to 8 h. Score ranges for SPID(0-4h), SPID(0-6), SPID(0-12) and SPID(0-24) are -12 to 4, -18 to 6, -36 to 12 and -72 to 24 respectively. Participants were required to have moderate (score=2) or severe (score=3) pain at baseline in order to be eligible for randomization.LS mean were calculated using ANCOVA and was adjusted for treatment as a fixed effect and baseline pain intensity as a continuous covariate. The measure of dispersion reported is 95% CrI not CI. A negative direction indicated a pain reduction from baseline.
  There were no planned efficacy analysis for Pre-Part B per protocol.
Time Frame: 0 to 4, 0 to 6, 0 to 8, 0 to 12, and 0 to 24 h post-dose
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Part A - LY3023703 | Part A - Celecoxib | Part A - Placebo | Part B - LY3023703 | Part B - Placebo
Number analyzed (Participants) | 30 | 31 | 30 | 15 | 15
units on a scale
  0 to 4 h | -0.6 [-1.5 to 0.3] | -4.1 [-5.0 to -3.2] | -1.2 [-2.1 to -0.3] | 0.0 [-0.9 to 1.0] | 0.3 [-0.6 to 1.3]
  0 to 6 h | -1.0 [-2.5 to 0.5] | -6.9 [-8.4 to -5.5] | -2.1 [-3.6 to -0.7] | 0.2 [-1.4 to 1.7] | 0.2 [-1.3 to 1.8]
  0 to 8 h | -1.3 [-3.4 to 0.7] | -9.4 [-11.4 to -7.3] | -3.2 [-5.3 to -1.2] | 0.3 [-1.9 to 2.5] | 0.1 [-2.1 to 2.4]
  0 to 12 h | -2.1 [-5.4 to 1.2] | -13.7 [-17.1 to -10.4] | -5.5 [-8.8 to -2.2] | 0.7 [-2.8 to 4.2] | -0.2 [-3.6 to 3.2]
  0 to 24 h | -5.2 [-12.5 to 2.4] | -27.1 [-34.4 to -19.8] | -13.0 [-20.2 to -5.6] | 2.4 [-5.4 to 10.1] | -1.7 [-9.4 to 5.9]
Statistical Analysis 1: Comparison: Part A - LY3023703 vs Part A - Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [-0.6 to 1.9] — 95% CrI is reported here, not the CI. Estimation is SPID 0 to 4 h
Statistical Analysis 2: Comparison: Part A - Celecoxib vs Part A - Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = -2.9, 95% CI 2-sided [-4.1 to -1.7] — 95% CrI is reported here, not the CI. Estimation is for SPID 0 to 4 h
Statistical Analysis 3: Comparison: Part A - LY3023703 vs Part A - Celecoxib; Test type: Superiority or Other; Mean Difference (Final Values) = 3.5, 95% CI 2-sided [2.3 to 4.8] — 95% CrI is reported here, not the CI. Estimation is for SPID 0 to 4 h
Statistical Analysis 4: Comparison: Part A - LY3023703 vs Part A - Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = 1.1, 95% CI 2-sided [-0.9 to 3.2] — 95% CrI is reported here, not the CI. Estimation is for SPID 0 to 6 h
Statistical Analysis 5: Comparison: Part A - Celecoxib vs Part A - Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = -4.8, 95% CI 2-sided [-6.8 to -2.7] — 95% CrI is reported here, not the CI. Estimation is for SPID 0 to 6 h
Statistical Analysis 6: Comparison: Part A - LY3023703 vs Part A - Celecoxib; Test type: Superiority or Other; Mean Difference (Final Values) = 5.9, 95% CI 2-sided [3.8 to 8.0] — 95% CrI is reported here, not the CI. Estimation is for SPID 0 to 6 h
Statistical Analysis 7: Comparison: Part A - LY3023703 vs Part A - Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = 1.9, 95% CI 2-sided [-1.0 to 4.8] — 95% CrI is reported here, not the CI. Estimation is for SPID 0 to 8 h
Statistical Analysis 8: Comparison: Part A - Celecoxib vs Part A - Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = -6.1, 95% CI 2-sided [-9.0 to -3.3] — 95% CrI is reported here, not the CI. Estimation is for SPID 0 to 8 h
Statistical Analysis 9: Comparison: Part A - LY3023703 vs Part A - Celecoxib; Test type: Superiority or Other; Mean Difference (Final Values) = 8.0, 95% CI 2-sided [5.1 to 10.9] — 95% CrI is reported here, not the CI. Estimation is for SPID 0 to 8 h
Statistical Analysis 10: Comparison: Part A - LY3023703 vs Part A - Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = 3.4, 95% CI 2-sided [-1.3 to 8.1] — 95% CrI is reported here, not the CI. Estimation is for SPID 0 to 12 h
Statistical Analysis 11: Comparison: Part A - Celecoxib vs Part A - Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = -8.2, 95% CI 2-sided [-12.9 to -3.5] — 95% CrI is reported here, not the CI. Estimation is for SPID 0 to 12 h
Statistical Analysis 12: Comparison: Part A - LY3023703 vs Part A - Celecoxib; Test type: Superiority or Other; Mean Difference (Final Values) = 11.6, 95% CI 2-sided [7.0 to 16.5] — 95% CrI is reported here, not the CI. Estimation is for SPID 0 to 12 h
Statistical Analysis 13: Comparison: Part A - LY3023703 vs Part A - Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = 7.8, 95% CI 2-sided [-2.6 to 18.3] — 95% CrI is reported here, not the CI. Estimation is for SPID 0 to 24 h
Statistical Analysis 14: Comparison: Part A - Celecoxib vs Part A - Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = -14.1, 95% CI 2-sided [-24.7 to -3.6] — 95% CrI is reported here, not the CI. Estimation is for SPID 0 to 24 h
Statistical Analysis 15: Comparison: Part A - LY3023703 vs Part A - Celecoxib; Test type: Superiority or Other; Mean Difference (Final Values) = 21.9, 95% CI 2-sided [11.5 to 32.2] — 95% CrI is reported here, not the CI. Estimation is for SPID 0 to 24 h
Statistical Analysis 16: Comparison: Part B - LY3023703 vs Part B - Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-1.6 to 1.0] — 95% CrI is reported here, not the CI. Estimation is for SPID 0 to 4 h
Statistical Analysis 17: Comparison: Part B - LY3023703 vs Part B - Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = -0.0, 95% CI 2-sided [-2.2 to 2.1] — 95% CrI is reported here, not the CI. Estimation is for SPID 0 to 6 h
Statistical Analysis 18: Comparison: Part B - LY3023703 vs Part B - Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-2.9 to 3.3] — 95% CrI is reported here, not the CI. Estimation is for SPID 0 to 8 h
Statistical Analysis 19: Comparison: Part B - LY3023703 vs Part B - Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = 0.9, 95% CI 2-sided [-3.9 to 5.7] — 95% CrI is reported here, not the CI. Estimation is for SPID 0 to 12 h
Statistical Analysis 20: Comparison: Part B - LY3023703 vs Part B - Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = 4.1, 95% CI 2-sided [-6.8 to 15.0] — 95% CrI is reported here, not the CI. Estimation is for SPID 0 to 24 h

5. Secondary Outcome: Time to First Use of Rescue Medication
Description: Time to first use of rescue medication is defined as the time from study drug administration to the measured first use of rescue medication in hours. Participants were censored at 24 h post-dose if no rescue medication was administered.
  Pre-Part B used 3 participants in order for the study site to develop proficiency in the dialysate placement, collection, and maintenance techniques. There were no planned efficacy analysis for Pre-Part B per protocol.
Time Frame: Study drug administration to first use of rescue medication (0 to 24 h post-dose)
Population: FAS: All data from all participants randomly assigned to treatment who received at least 1 dose of study medication and who had at least 1 post-dose efficacy assessment. Participants censored: Part A: LY3023703=5, Celecoxib=18, Placebo=12, Part B: LY3023703=0, Placebo=2.
Measure: Median (95% Confidence Interval); unit: h
Arm/Group | Part A - LY3023703 | Part A - Celecoxib | Part A - Placebo | Part B - LY3023703 | Part B - Placebo
Number analyzed (Participants) | 30 | 31 | 30 | 15 | 15
h | 1.8 [1.7 to 2.3] | NA [8.3 to NA] — Median and upper limit of CI were not calculated, less than 50% of participants received rescue medication. | 2.9 [1.8 to NA] — Upper limit of CI was not calculated, less than 50% of participants received rescue medication. | 1.9 [1.7 to 1.9] | 1.8 [1.8 to 2.2]
Statistical Analysis 1: Comparison: Part A - LY3023703 vs Part A - Placebo; Test type: Superiority or Other; Cox Proportional Hazard = 1.85, 95% CI 2-sided [0.99 to 3.46] — Hazard ratio (HR) of the treatment differences were estimated based on Cox proportional hazard model including treatment and baseline pain intensity (VAS) as fixed effects
Statistical Analysis 2: Comparison: Part A - Celecoxib vs Part A - Placebo; Test type: Superiority or Other; Cox Proportional Hazard = 0.34, 95% CI 2-sided [0.16 to 0.72] — HR of the treatment differences were estimated based on Cox proportional hazard model including treatment and baseline pain intensity (VAS) as fixed effects
Statistical Analysis 3: Comparison: Part A - LY3023703 vs Part A - Celecoxib; Test type: Superiority or Other; Cox Proportional Hazard = 5.48, 95% CI 2-sided [2.69 to 11.16] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 4: Comparison: Part B - LY3023703 vs Part B - Placebo; Test type: Superiority or Other; Cox Proportional Hazard = 1.22, 95% CI 2-sided [0.57 to 2.59] — [estimate comment as in outcome 5, analysis 2]

6. Secondary Outcome: Part A: Time to Onset of First Perceptible Pain Relief
Description: Time to onset of the first perceptible pain relief is defined as the time from study drug administration to the measured onset of first perceptible pain relief in hours as reported by the participant. Participants who received rescue mediation prior to first perceptible pain relief were censored at the time the rescue medication was received.
Time Frame: Study drug administration to first perceptible pain relief (0 to 24 h post-dose)
Population: FAS: Part A participants randomly assigned to treatment who received at least 1 dose of study medication and who had at least 1 post-dose efficacy assessment. Participants censored: Part A: LY3023703=11, Celecoxib=2, Placebo=9.
Measure: Median (95% Confidence Interval); unit: h
Arm/Group | Part A - LY3023703 | Part A - Celecoxib | Part A - Placebo
Number analyzed (Participants) | 30 | 31 | 30
h | 0.9 [0.6 to 2.2] | 0.7 [0.4 to 0.8] | 1.0 [0.4 to 1.6]
Statistical Analysis 1: Comparison: Part A - LY3023703 vs Part A - Placebo; Test type: Superiority or Other; Cox Proportional Hazard = 0.78, 95% CI 2-sided [0.41 to 1.47] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 2: Comparison: Part A - Celecoxib vs Part A - Placebo; Test type: Superiority or Other; Cox Proportional Hazard = 2.15, 95% CI 2-sided [1.19 to 3.88] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 3: Comparison: Part A - LY3023703 vs Part A - Celecoxib; Test type: Superiority or Other; Cox Proportional Hazard = 0.36, 95% CI 2-sided [0.19 to 0.67] — [estimate comment as in outcome 5, analysis 2]

7. Secondary Outcome: Part A: Time to Onset of Meaningful Pain Relief
Description: Time to onset of meaningful pain relief is defined as the time from study drug administration to the measured onset of meaningful pain relief in hours as reported by the participant. Participants who received rescue mediation prior to meaningful pain relief were censored at the time the rescue medication was received.
Time Frame: Study drug administration to meaningful pain relief (0 to 24 h post-dose)
Population: FAS: Part A participants randomly assigned to treatment who received at least 1 dose of study medication and who had at least 1 post-dose efficacy assessment. Participants censored: Part A LY3023703=24, Celecoxib=2, Placebo=15.
Measure: Median (95% Confidence Interval); unit: h
Arm/Group | Part A - LY3023703 | Part A - Celecoxib | Part A - Placebo
Number analyzed (Participants) | 30 | 31 | 29
h | 3.8 [3.0 to 3.8] | 1.2 [0.9 to 1.4] | 2.2 [1.6 to 4.9]
Statistical Analysis 1: Comparison: Part A - LY3023703 vs Part A - Placebo; Test type: Superiority or Other; Cox Proportional Hazard = 0.33, 95% CI 2-sided [0.12 to 0.88] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 2: Comparison: Part A - Celecoxib vs Part A - Placebo; Test type: Superiority or Other; Cox Proportional Hazard = 4.16, 95% CI 2-sided [2.04 to 8.47] — [estimate comment as in outcome 5, analysis 2]
Statistical Analysis 3: Comparison: Part A - LY3023703 vs Part A - Celecoxib; Test type: Superiority or Other; Cox Proportional Hazard = 0.08, 95% CI 2-sided [0.03 to 0.21] — [estimate comment as in outcome 5, analysis 2]

8. Secondary Outcome: Part A: Patient Global Impression of Improvement (PGI-I) Scale Score
Description: PGI-I is a participant-rated instrument that measures the improvement of the participants symptoms on a 7-point scale: 1 (very much improved), 4 (no change), and 7 (very much worse). LS mean was calculated using Mixed Effect Model Repeated Measures (MMRM) adjusted for treatment, time, the interaction of treatment and time and baseline pain VAS and fixed effects.
Time Frame: 2, 4, 8, 12 and 24 h post-dose
Population: Part A participants who were randomly assigned to treatment who received at least 1 dose of study medication and who had at least 1 post-dose PGI-I assessment. Participants who received rescue medication were not included in the specific timepoints post administration of rescue medication.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Part A - LY3023703 | Part A - Celecoxib | Part A - Placebo
Number analyzed (Participants) | 10 | 29 | 19
units on a scale
  2 h | 2.91 [2.41 to 3.41] | 1.95 [1.65 to 2.25] | 3.12 [2.75 to 3.49]
  4 h: number analyzed (Participants) | 5 | 29 | 12
  4 h | 2.17 [1.68 to 2.67] | 1.92 [1.68 to 2.16] | 2.45 [2.12 to 2.78]
  8 h: number analyzed (Participants) | 5 | 22 | 12
  8 h | 2.29 [1.66 to 2.92] | 1.96 [1.66 to 2.26] | 1.94 [1.53 to 2.34]
  12 h: number analyzed (Participants) | 5 | 19 | 12
  12 h | 1.91 [1.22 to 2.59] | 2.03 [1.70 to 2.37] | 1.78 [1.34 to 2.23]
  24 h: number analyzed (Participants) | 5 | 18 | 12
  24 h | 1.29 [0.81 to 1.76] | 1.74 [1.50 to 1.98] | 1.34 [1.03 to 1.65]

ADVERSE EVENTS:
Arm/Group | Part A - LY3023703 | Part A - Celecoxib | Part A - Placebo | Part B - LY3023703 | Part B - Placebo | Pre-Part B - Celecoxib
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/31 | 0/30 | 0/15 | 0/15 | 0/3
Other Adverse Events (participants affected / at risk) | 4/30 | 4/31 | 6/30 | 4/15 | 8/15 | 0/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A - LY3023703 (N=30) | Part A - Celecoxib (N=31) | Part A - Placebo (N=30) | Part B - LY3023703 (N=15) | Part B - Placebo (N=15) | Pre-Part B - Celecoxib (N=3)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site bruise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alveolar osteitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 4 (4) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Body temperature increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Papule (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days